CLINICAL TRIAL: NCT04335565
Title: Effect of Stevia Extract on Postprandial Glucose Response and Satiety in Overweight and Obese Adults: A Three-arm Crossover Trial.
Brief Title: Stevia Extract and Glucose Homeostasis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been terminated due to the pandemic.
Sponsor: Liverpool Hope University (Other)
Responsible Party: Principal Investigator, Grace Farhat, Dr, Liverpool Hope University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 13022020
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-04

CONDITIONS: Overweight; Obesity
Keywords: Non-nutritive sweeteners; postprandial glucose; diabetes; obesity; satiety
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water (No Intervention): 250 ml of water mixed with 1g of citric acid.
- Sugar (Active Comparator): 65g of sugar dissolved in 250ml of water
  Interventions: Other: sugar replacements
- Stevia (Experimental): 5g of stevia dissolved in 250ml of water
  Interventions: Other: sugar replacements

INTERVENTIONS:
Other: sugar replacements — Participants will receive a solution of stevia before being administered a fixed meal (lunch). Glucose and insulin levels, and Visual analogue scale data will be collected.
  Arms: Stevia; Sugar

SUMMARY:
This study aims to assess the effect of stevia extract on postprandial glucose and insulin levels in overweight and obese adults when compared to sugar and water.

DETAILED DESCRIPTION:
The study is a three-arm crossover trial involving participants attending the Lab on 3 different occasions (separated by 3-5 day washout period), where they will be administered water, sugar solution (65g), water and stevia extract (5g) solution. The solution will be followed by a consumption of a fixed meal (after 30 minutes). Breakfast will be standardised. Capillary blood glucose will be collected every 30 min until 2 hours post meal. Venous blood samples will be collected before the intake of the solution and at 2 hours after meal intake.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* BMI 27-40 Kg/m2
* Males and females

Exclusion Criteria:

* Athletes
* Pregnant or breastfeeding women
* Patients with chronic disease (diabetes, CVD etc…).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose levels | Capillary blood glucose will be measured two hours after the administration of a fixed meal.
  Change in glucose levels two hours after the administration of a fixed meal

SECONDARY OUTCOMES:
Postprandial insulin levels | Postprandial insulin levels will be measured two hours of the administration of a fixed meal
  Change in postprandial insulin levels two hours after the administration of a fixed meal
Area under the curve (AUC) for glucose | Capillary blood glucose levels will be collected 6 times on each visit before the intake of the solution until 2 hours post lunch
  Changes in AUC for glucose throughout the intervention
Subjective feelings of satiety | VAS will be collected 6 times on each visit before the intake of the solution until 2 hours post lunch.
  Visual analogue scales

CONTACTS AND LOCATIONS:
Overall Officials: Farzad Amirabdollahian, PhD, Study Chair — Liverpool Hope University
Locations (1):
- School of Health sciences, Liverpool Hope University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farhat G, Berset V, Moore L. Effects of Stevia Extract on Postprandial Glucose Response, Satiety and Energy Intake: A Three-Arm Crossover Trial. Nutrients. 2019 Dec 12;11(12):3036. doi: 10.3390/nu11123036. PMID 31842388